CLINICAL TRIAL: NCT02759835
Title: A Pilot Study of Local Ablative Therapy for Treatment of Oligoprogressive, EGFR-mutated, Non-Small Cell Lung Cancer (NSCLC) After Treatment With Osimertinib (AZD9291, Tagrisso)
Brief Title: Local Ablative Therapy for Treatment of Oligoprogressive, EGFR-Mutated, Non-Small Cell Lung Cancer After Treatment With Osimertinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Azam Ghafoor, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160092; 16-C-0092
Record Dates: First submitted 2016-04-06; First posted 2016-05-03 (Estimated); Results first posted 2023-07-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Lung Adenocarcinoma; Lung Neoplasms
Keywords: EGFR Tyrosine Kinase Inhibitors; T790M Mutation; Local Ablative Therapies; Oligoprogressive Disease; Acquired Resistance
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *mutated Non Small Cell Lung Cancer (Experimental): Cohort 1 - Osimertinib followed by LAT followed by osimertinib. Single daily dose of osimertinib until progression. The starting dose of osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline.
  *including germline T790M mutation
  Interventions: Drug: osimertinib; Other: Local Ablative Therapy (LAT)
- EGFR mutated NSCLC Progressed on prior 1st/2nd Generation EGFR TKI therapy &acquired T790M Mutation (Experimental): Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation.
  Interventions: Drug: osimertinib; Other: Local Ablative Therapy (LAT)
- Epidermal Growth Factor Receptor mutated Non Small Cell Lung Cancer Progressed on Osimertinib (Experimental): Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Interventions: Drug: osimertinib; Other: Local Ablative Therapy (LAT)

INTERVENTIONS:
Drug: osimertinib — Single daily dose of osimertinib until progression. The starting dose of osimertinib will be 80 mg per day for patients without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline.
  Other Names: Tagrisso
Other: Local Ablative Therapy (LAT) — local ablative therapy. Subjects may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, radiofrequency ablation

SUMMARY:
Background:

Some non-small-cell lung cancers (NSCLC) have a mutation in a gene that makes a protein called EGFR. This particular cancer can be treated with certain drugs such as erlotinib (Tarceva), gefitinib (Iressa) and osimertinib (Tagrisso). But many tumors become resistant to these drugs because of a second mutation. Researchers want to test if adding local ablative therapy (LAT) extends the benefits of the drug, osimertinib. LAT can include techniques such as surgery, radiofrequency ablation, cryotherapy or radiation therapy.

Objective:

To test if re-taking osimertinib after LAT is safe, tolerable, and effective for people whose NSCLC has progressed after initial treatment with osimertinib.

Eligibility:

Adults ages 18 and older with certain types of NSCLC. Participants will be divided into various groups as described below.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Tumor scans

Eye exam

Review of tumor sample.

Participants will take the study drug by mouth once a day. They will continue until they can no longer tolerate it or their disease worsens. They will keep a dosage diary.

All participants will start each 21-day course with physical exam; blood, urine, and saliva tests; and electrocardiogram. They will have scans every 6 weeks and echocardiogram every 3 months.

Groups 1 and 2 will:

Start osimertinib right away.

Have LAT if their disease progresses and is suitable for LAT. If LAT cannot be performed or LAT consists of a procedure other than surgery, a tumor biopsy will be performed.

Re-start osimertinib after LAT, or other treatments if not suitable for LAT.

Group 3 will:

Have LAT.

If LAT consists of a procedure other than surgery, a tumor biopsy will be performed.

Start osimertinib after LAT.

After participants stop taking the drugs, they will have a final visit. This will include:

Medical history

Physical exam

Blood tests

Participants will be called every year for follow-up.

DETAILED DESCRIPTION:
Background:

* Epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKI) have significantly improved the response rate (RR) and survival in patients with tumors harboring EGFR-sensitizing mutations.
* An invariable consequence of treatment with EGFR-TKIs is the development of acquired resistance. The most common mechanism of resistance observed in approximately 50% of all cases in patients treated with 1st and 2nd generation EGFR-TKIs is the emergence of a secondary mutation (T790M) in exon 20.
* Osimertinib is a 3rd-generation EGFR-TKI designed to target the T790M mutation, which has shown impressive responses in both first- and second-line settings.
* Despite these developments, it is almost certain that selection pressure will lead to the emergence of newer clones that are resistant to treatment with osimertinib. One common mechanism of acquired resistance to osimertinib is the generation of EGFR C797S mutation.
* The use of local ablative therapies for patients who develop limited metastatic disease or oligoprogressive disease on EGFR-TKI therapy is promising.
* We hypothesize that following local ablative therapy to treat oligoprogressive disease after emergence of resistance, osimertinib can be resumed safely and re-initiation of osimertinib results in additional progression-free survival benefits.

Objectives:

* Determine the safety, tolerability, and efficacy (as assessed by progression free survival (PFS) upon re-initiation of osimertinib following local ablative therapy (LAT) for patients with oligoprogressive disease after treatment with osimertinib
* Assess mechanisms of acquired resistance to osimertinib

Eligibility:

* Histologically confirmed advanced lung adenocarcinoma with EGFR-sensitizing somatic mutations or a germline T790M mutation and no prior EGFR tyrosine kinase inhibitor (TKI) therapy (Cohort 1); OR progressive disease after 1st or 2nd generation EGFR TKI therapy harboring somatic T790M mutation (Cohort 2); or patients with progressive disease after treatment with osimertinib who are eligible for local ablative therapy (Cohort 3). If biopsy for EGFR mutation status confirmation is not clinically feasible, EGFR mutations may be confirmed by circulating tumor deoxyribonucleic acid (ctDNA) analysis using a Clinical Laboratory Improvement Amendments of 1988 (CLIA) certified assay.
* Presence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate end organ function
* If patients are not eligible for LAT, they will be referred for standard of care chemotherapy as per treating physician's discretion. These patients may also be considered for other clinical trials.

Design:

* This is a single-institution, open-label phase II trial of osimertinib treatment in EGFR mutant lung cancer.
* Eligible patients not previously treated with osimertinib will be treated with osimertinib daily until disease progression. At the time of progression, patients with oligoprogressive disease (no more than 5 sites of progressive disease) will be assessed for LAT.
* If patients are eligible for LAT, osimertinib will be resumed after LAT and they will be followed for second progression on osimertinib (PFS2).
* If patients progress at the same site where LAT has been performed before, the progression will be considered to be a result of inadequate ablation and they will be considered for repeat LAT and again re-challenged with osimertinib if clinically feasible.
* Tumor samples will be obtained at baseline by a mandatory biopsy. At the time of first progression on osimertinib if a patient is eligible for surgery as a form of LAT, then a tissue sample will be obtained for genomic and proteomic studies to identify mechanisms of acquired resistance. For patients who are not eligible for LAT or a form of LAT that is not surgery (radiation, radiofrequency ablation, cryoablation), then a mandatory biopsy will be performed, if clinically safe, to obtain tissue for above studies.
* Re-treatment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

For inclusion in the study subjects should fulfill the following criteria:

* Provision of informed consent prior to any study specific procedures
* Patients (male/female) must be greater than or equal to 18 years of age.
* Patients with histologically confirmed, by the National Cancer Institute (NCI) Laboratory of Pathology or by Clinical Laboratory Improvement Amendments of 1988 (CLIA)-certified Next Generation Sequencing or Cobas estimated Epidermal Growth Factor Receptor (EGFR) Mutation Test v1/2 at an outside institution, advanced lung adenocarcinoma with EGFR-sensitizing somatic mutations or a germline T790M mutation (detected histologically or via circulating tumor deoxyribonucleic acid (ctDNA) analysis using a CLIA assay) with:

  * No prior EGFR tyrosine kinase inhibitor (TKI) therapy (Cohort 1)

OR

-- Progressive disease after 1st or 2nd generation EGFR TKI therapy harboring somatic T790M mutation (Cohort 2)

OR

* Progressive disease after treatment with osimertinib who are eligible for local ablative therapy (Cohort 3)

  * Presence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  * In patients with suspected leptomeningeal disease, the diagnosis of leptomeningeal disease should be confirmed by the presence of neurological or imaging signs and/or positive cerebrospinal fluid (CSF) cytology.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
  * No uncontrolled arrhythmia; no myocardial infarction in the last 6 months.
  * Females should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
* Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
* Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing Hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

  * Females of child-bearing potential should use reliable methods of contraception from the time of screening until 3 months after discontinuing osimertinib. Acceptable methods of contraception include total and true sexual abstinence, tubal ligation, hormonal contraceptives that are not prone to drug-drug interactions (IUS Levonorgestrel Intra Uterine System (Mirena), Medroxyprogesterone injections (Depo-Provera), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their male sexual partner for intercourse.
  * Male patients should be willing to use barrier contraception. Male patients should be asked to use barrier contraceptives (i.e., by use of condoms) during sex with all of their female partners during the trial and for a washout period of 3 months. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing osimertinib treatment. If male patients wish to father children, they should be advised to arrange for freezing of sperm samples prior to the start of osimertinib treatment.
  * Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

EXCLUSION CRITERIA:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception, of alopecia and grade 2, prior platinum-therapy related neuropathy.
* Treatment with an investigational drug within five half-lives of the compound.
* Major thoracic or abdominal surgery from which the patient has not sufficiently recovered yet.
* Untreated and uncontrolled second tumor in the past 2 years.
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of cytochrome P450 3A4 (CYP3A4) (at least 3 weeks prior) will only be eligible at the PI's discretion.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
* Patients with central nervous system (CNS) metastases who are neurologically unstable.
* Past medical history of interstitial lung disease (ILD), drug induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count <1 x 10(9)/L
  * Platelet count <100 x 10(9)/L
  * Hemoglobin <90 g/L
  * Alanine aminotransferase >2.5 times the 2.1.2.9.4 upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
  * Creatinine >1.5 times ULN concurrent with creatinine clearance <30 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
* Any of the following cardiac criteria

  * Resting corrected QT interval (corrected QT interval (QTc) using Fredericia's formula) > 480 msec
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
  * Significant symptomatic congestive heart failure, per principal investigator (PI) judgement.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
* History of hypersensitivity to osimertinib (or drugs with a similar chemical structure or class to osimertinib) or any excipients of these agents
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azam Ghafoor, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing Plan (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Result] Kim C, Xi L, Cultraro CM, Wei F, Jones G, Cheng J, Shafiei A, Pham TH, Roper N, Akoth E, Ghafoor A, Misra V, Monkash N, Strom C, Tu M, Liao W, Chia D, Morris C, Steinberg SM, Bagheri H, Wong DTW, Raffeld M, Guha U. Longitudinal Circulating Tumor DNA Analysis in Blood and Saliva for Prediction of Response to Osimertinib and Disease Progression in EGFR-Mutant Lung Adenocarcinoma. Cancers (Basel). 2021 Jul 3;13(13):3342. doi: 10.3390/cancers13133342. PMID 34283064
- [Result] Roper N, Brown AL, Wei JS, Pack S, Trindade C, Kim C, Restifo O, Gao S, Sindiri S, Mehrabadi F, El Meskini R, Ohler ZW, Maity TK, Venugopalan A, Cultraro CM, Akoth E, Padiernos E, Chen H, Kesarwala A, Smart DK, Nilubol N, Rajan A, Piotrowska Z, Xi L, Raffeld M, Panchenko AR, Sahinalp C, Hewitt S, Hoang CD, Khan J, Guha U. Clonal Evolution and Heterogeneity of Osimertinib Acquired Resistance Mechanisms in EGFR Mutant Lung Cancer. Cell Rep Med. 2020 Apr 21;1(1):100007. doi: 10.1016/j.xcrm.2020.100007. PMID 32483558
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0092.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
- EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
Period: Overall Study
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Started | 25 | 9 | 3
Completed | 25 | 9 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib | Total
Number analyzed (Participants) | 25 | 9 | 3 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 5 | 3 | 22
  >=65 years | 11 | 4 | 0 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.54 (15.03) | 58.86 (11.48) | 60.13 (3.91) | 59.67 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 3 | 27
  Male | 8 | 2 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 23 | 8 | 2 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 0 | 1 | 9
  White | 9 | 6 | 1 | 16
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 9 | 3 | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival 1 (PFS 1) for ALL Participants Who Started Osimertinib on Trial Until First Progression of Disease or Clinical Progression, or Death Any Cause
Description: PFS1 = time from initiation of osimertinib to first progression of disease or clinical progression, or death any cause. Progression was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and reported using the Kaplan Meier curve. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progression).
Time Frame: Cycle 1 Day 1 (each cycle is 28 days) to progression of disease, range 36-1231 days
Population: Cohort 3 is not applicable for this outcome measure because these participants enrolled in the study after getting Osimertinib at an outside institution. One participant in Cohort 1 was not evaluable.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants in Cohort 1: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
- All Participants in Cohort 2: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
Arm/Group | All Participants in Cohort 1 | All Participants in Cohort 2
Number analyzed (Participants) | 24 | 9
Months | 14.7 [5.6 to 22.0] | 11.0 [5.5 to 25.7]
Statistical Analysis 1: Comparison: All Participants in Cohort 1 vs All Participants in Cohort 2; Test type: Other; p = 0.56, Kaplan-Meier

2. Primary Outcome: Progression Free Survival 2 (PFS 2) - Local Ablative Therapy (LAT Eligible Only)
Description: PFS2 = time from osimertinib re-challenge after LAT following first progression on osimertinib until second progression on osimertinib. Progression was evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and reported using the Kaplan Meier curve. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progression).
Time Frame: Retreatment Cycle 1 Day 1 (cycle is 28 days) to progression of disease, range 29-721 days
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants in Cohorts 1, 2, and 3: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
Arm/Group | All Participants in Cohorts 1, 2, and 3
Number analyzed (Participants) | 21
Months | 3.7 [1.9 to 4.6]

3. Primary Outcome: Progression Free Survival 2 (PFS 2) - Local Ablative Therapy (LAT Eligible Only) - Cohort 1, Cohort 2, and Cohort 3
Description: as for outcome 2
Time Frame: Retreatment Cycle 1 Day 1 (cycle is 28 days) to progression of disease, range 29-721 days
Population: This outcome measure reports data for LAT eligible participants only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 12 | 6 | 3
Months | 4.0 [1.0 to 16.5] | 3.6 [1.8 to 4.6] | 3.7 [2.3 to 23.9]
Statistical Analysis 1: Comparison: Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer vs EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation vs Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib; Test type: Other; p = 0.40, Kaplan-Meier

4. Primary Outcome: Serious Adverse Events Possibly, Probably, and/or Definitely Related to Treatment
Description: Adverse events were assessed by the by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 74 months and 16 days, 65 months and 16 days, and 40 months and 4 days for the first, second and third group respectively.
Measure: Number; unit: adverse events
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 25 | 9 | 3
adverse events
  Anemia - Possibly Related | 1 | 0 | 0
  Lung Infection - Possibly Related | 1 | 0 | 0
  Peripheral Sensory Neuropathy Possibly Related | 1 | 0 | 0
  Pleural Effusion - Possibly Related | 1 | 0 | 0
  Thromboembolic Event - Definitely Related | 1 | 0 | 0

5. Primary Outcome: All Grades 1, Grade 2, Grade 3, Grade 4, and/or Grade 5 Adverse Events Possibly, Probably, and/or Definitely Related to Local Ablative Therapy (LAT)
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse events.
Time Frame: as for outcome 4
Measure: Number; unit: adverse events
Groups:
- Cohort 1: Possibly Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Adverse events possibly related to LAT.
- Cohort 1: Probably Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Adverse events probably related to LAT.
- Cohort 1: Definitely Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation.
  Adverse events definitely related to LAT.
- Cohort 2: Possibly Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events possibly related to LAT.
- Cohort 2: Probably Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events probably related to LAT.
- Cohort 2: Definitely Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events definitely related to LAT.
- Cohort 3: Possibly Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events possibly related to LAT.
- Cohort 3: Probably Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events probably related to LAT.
- Cohort 3: Definitely Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events definitely related to LAT.
Arm/Group | Cohort 1: Possibly Related | Cohort 1: Probably Related | Cohort 1: Definitely Related | Cohort 2: Possibly Related | Cohort 2: Probably Related | Cohort 2: Definitely Related | Cohort 3: Possibly Related | Cohort 3: Probably Related | Cohort 3: Definitely Related
Number analyzed (Participants) | 25 | 25 | 25 | 9 | 9 | 9 | 3 | 3 | 3
adverse events
  Abdominal pain - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase - increased - Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase - increased - Grade 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased - Grade 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia -Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia - Grade 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Arthralgia - Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Atelectasis - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bloating - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blurred vision - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CPK increased - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cough - Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cough - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness - Grade 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Dry mouth - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dysgeusia - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea - Grade 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Dyspnea - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram QT corrected interval prolonged - Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Eyelid function disorder - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fall - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fever - Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia - Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia - Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypotension - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypotension - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoxia - Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Localized edema - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle weakness upper limb - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Muscle weakness lower limb - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle weakness lower limb - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea - Grade 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Non-cardiac chest pain - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Non-cardiac chest pain - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pain - Grade 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Pain - Grade 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pain - Grade 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Pain in extremity - Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paresthesia - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pericardial effusion - Grade 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Peripheral sensory neuropathy - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pleural effusion - Grade 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pleural effusion - Grade 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Pleural effusion - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pneumothorax - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pneumothorax - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Other, Hydropneumothorax - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Hydropneumothorax - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Other, Subcutaneous emphysema - Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Sore throat - Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Sinus tachycardia - Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Surgical and medical procedures - Other, incision site pain - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Surgical and medical procedures - Other, incision site pain - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tinnitus - Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinary retention - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting - Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Wheezing - Grade 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Wheezing - Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: All Grades 1, Grade 2, Grade 3, Grade 4, and/or Grade 5 Adverse Events Possibly, Probably, and/or Definitely Related to Osimertinib
Description: as for outcome 5
Time Frame: as for outcome 4
Population: *Because this adverse event has attribution to local ablative therapy (LAT) as well.
Measure: Number; unit: adverse events
Groups:
- Cohort 1: Possibly Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Adverse events possibly related to osimertinib.
- Cohort 1: Probably Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Adverse events probably related to osimertinib.
- Cohort 1: Definitely Related: COHORT 1: Osimertinib followed by LAT followed by osimertinib. Single daily dose of Osimertinib until progression. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation.
  *including germline T790M mutation
  Adverse events definitely related to osimertinib.
- Cohort 2: Possibly Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events possibly related to osimertinib.
- Cohort 2: Probably Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events probably related to osimertinib.
- Cohort 2: Definitely Related: Cohort 2 - Osimertinib followed by LAT followed by osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on osimertinib: surgery, radiotherapy, or radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events definitely related to osimertinib.
- Cohort 3: Possibly Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events possibly related to osimertinib.
- Cohort 3: Probably Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events probably related to osimertinib.
- Cohort 3: Definitely Related: Cohort 3 - LAT followed by Osimertinib. Participants may undergo 1 of 3 local ablative procedures after initial progression on Osimertinib: surgery, radiotherapy, radiofrequency ablation. The starting dose of Osimertinib will be 80 mg per day for participants without leptomeningeal disease and 160 mg per day for those with leptomeningeal disease at baseline. Single daily dose of Osimertinib until progression.
  Adverse events definitely related to osimertinib.
Arm/Group | Cohort 1: Possibly Related | Cohort 1: Probably Related | Cohort 1: Definitely Related | Cohort 2: Possibly Related | Cohort 2: Probably Related | Cohort 2: Definitely Related | Cohort 3: Possibly Related | Cohort 3: Probably Related | Cohort 3: Definitely Related
Number analyzed (Participants) | 25 | 25 | 25 | 9 | 9 | 9 | 3 | 3 | 3
adverse events
  Alanine aminotransferase increased - Grade 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alopecia - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia - Grade 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Anemia - Grade 1* | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia - Grade 2 | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Anemia - Grade 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia - Grade 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia - Grade 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bloating - Grade 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blurred vision - Grade 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blurred vision - Grade 1* | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Buttock pain - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CPK increased - Grade 1 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CPK increased - Grade 2 | 5 | 4 | 0 | 7 | 0 | 0 | 0 | 0 | 0
  CPK increased - Grade 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CPK increased - Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Constipation - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cough - Grade 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea - Grade 1 | 4 | 6 | 4 | 4 | 2 | 0 | 1 | 0 | 0
  Diarrhea - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Dizziness - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry eye - Grade 1 | 3 | 4 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Dry mouth - Grade 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry skin - Grade 1 | 9 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0
  Dry skin - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
  Dysgeusia - Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspepsia - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Dyspepsia - Grade 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Dyspnea - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema face - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema limbs - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram QT corrected interval prolonged - Grade 1 | 9 | 2 | 0 | 12 | 5 | 0 | 1 | 0 | 0
  Electrocardiogram QT corrected interval prolonged - Grade 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Electrocardiogram QT corrected interval prolonged - Grade 2* | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Esophagitis - Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye pain - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue - Grade 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  Fatigue - Grade 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Floaters - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastritis - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastroesophageal reflux disease - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Gastroesophageal reflux disease - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Other, stomatitis - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Other, stomatitis - Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Headache - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Headache - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypertension - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia - Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypophosphatemia - Grade 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lung infection - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 1 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Lymphocyte count decreased - Grade 2* | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 3 | 19 | 1 | 0 | 4 | 1 | 0 | 2 | 0 | 0
  Lymphocyte count decreased - Grade 3* | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased - Grade 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Metabolism and nutrition disorders - Other, muscle cramps - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucositis oral - Grade 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucositis oral - Grade 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mucositis oral - Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia - Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nail infection - Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nail loss - Grade 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Nail loss - Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nail ridging - Grade 1 | 4 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Nausea - Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased - Grade 2 | 4 | 3 | 0 | 3 | 1 | 0 | 0 | 1 | 0
  Neutrophil count decreased - Grade 3 | 14 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Neutrophil count decreased - Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-cardiac chest pain - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain in extremity - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Palmar-plantar erythrodysesthesia syndrome - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Palmar-plantar erythrodysesthesia syndrome - Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Papulopustular rash - Grade 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Papulopustular rash - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paronychia - Grade 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paronychia - Grade 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Peripheral sensory neuropathy - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Photophobia - Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased - Grade 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Platelet count decreased - Grade 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Platelet count decreased - Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Pleural effusion - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Productive cough -Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritis - Grade 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pruritis - Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Rash acneiform - Grade 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Rash acneiform - Grade 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Rash maculo-papular - Grade 1 | 12 | 7 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Rash maculo-papular - Grade 2 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Rash maculo-papular - Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Rash pustular - Grade 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Other, Cracks around fingertips - Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Crack right and left thumb and left 3rd finger - Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin hypopigmentation - Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Other, mild cracks at fingertips - Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Thromboembolic event - Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting - Grade 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Watering eyes - Grade 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Watering eyes - Grade 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight loss - Grade 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Weight loss - Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased - Grade 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  White blood cell decreased - Grade 2 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased - Grade 3 | 16 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Had Osimertinib Acquired Resistant Mechanisms Identified on Tumors
Description: Whole-exome sequencing (WES), targeted sequencing and ribonucleic acid (RNA)-seq was performed on tumors to identify Osimertinib acquired resistant mechanisms. Sequencing can help identify mutations/heterogeneity that may impact a participant prognosis.
Time Frame: up to 757 days
Population: 15/37 participants had tissue available for analysis and 2/37 participants were censored.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 9 | 3 | 3
Participants
  ≥1 resistance mechanisms | 9 | 3 | 3
  2 or more resistance mechanisms co-occurring | 8 | 2 | 2

8. Primary Outcome: Number of Participants Who Had Osimertinib Acquired Resistant Mechanisms Identified on Tumors With First Line and/or Second Line Treatment
Description: Whole-exome sequencing (WES), targeted sequencing and ribonucleic acid (RNA)-seq was performed on tumors for first and second line Osimertinib treatment to identify Osimertinib acquired resistant mechanisms. Sequencing can help identify mutations (i.e., NE-differentiation, ribonucleic acid (RNA), v-raf murine sarcoma viral oncogene homolog B1 (BRAF), other amps, etc.)/heterogeneity that may impact a participant prognosis.
Time Frame: up to 757 days
Population: 15/37 participants had tissue available for analysis and 2/37 participants were censored.
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 9 | 3 | 3
Participants
  Casitas B-lineage lymphoma(Cbl), Kirsten Rat Sarcoma(KRAS),MET&other amplification (amps)-First Line | 1 | 0 | 0
  mesenchymal epithelial transition factor receptor (MET) amps -First Line | 1 | 0 | 0
  Epidermal growth factor receptor (EGFR) amp & EGFR C797S mutation - Second Line | 0 | 1 | 0
  Small Cell Lung Cancer (SCLC) transformation - Second Line | 0 | 0 | 1
  Epidermal growth factor receptor (EGFR), MET amp & tumor protein P53 (TP53) A24fs -First Line | 1 | 0 | 0
  TP53 G112V & Catenin Beta 1(CTNNB1) Substitution-Missense,position 33, S➞C(S33C)mutations-First Line | 0 | 0 | 1
  Mixed Non-Small Cell Lung Cancer (NSCLC) & Small Cell Lung Cancer (SCLC) transformation - First Line | 1 | 0 | 0
  Unknown by exome; NE-differentiation without histologic transformation by RNA-seq-Second Line | 0 | 1 | 0
  Epidermal growth factor receptor (EGFR), Kirsten Rat Sarcoma (KRAS) & MET amp - First Line | 1 | 0 | 0
  mesenchymal epithelial transition factor receptor (MET) & other amps & EGFR C797S- Second Line | 1 | 0 | 1
  AGK(2) - BRAF(8) fusion & Makorin Ring Finger Protein 1 (MKRN1)(4) - BRAF(11) fusion - Second Line | 0 | 1 | 0
  Epidermal growth factor receptor (EGFR) & YES1 amp - Second Line | 1 | 0 | 0
  CD274 Programmed death-ligand 1 (PD-L1) & MET amp - First Line | 1 | 0 | 0
  Epidermal growth factor receptor(EGFR) C797S&estrogen receptor 1(ESR1(6)-AKAP12(4) fusion-First Line | 1 | 0 | 0
  Epidermal growth factor receptor(EGFR) & MET amp - First Line | 1 | 0 | 0

9. Secondary Outcome: Best Overall Response (BOR)
Description: Best Overall Response is defined as a Complete Response (CR) + Partial Response (PR) and is recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria. Response was evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions.
Time Frame: end of treatment, up to 693 days
Population: One participant was not evaluable for response in Cohort 1. Cohort 3 did not have a first treatment of Osimertinib on this protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 25 | 9 | 3
percentage of participants
  First Treatment - Complete Response + Partial Response: number analyzed (Participants) | 25 | 9 | 0
  First Treatment - Complete Response + Partial Response | 70.8 | 66.7 |
  Second Treatment - Complete Response + Partial Response | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Best Overall Response - All Participants
Description: as for outcome 9
Time Frame: end of treatment, up to 693 days
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | All Participants in Cohorts 1, 2, and 3
Number analyzed (Participants) | 36
percentage of participants
  First treatment - Complete Response + Partial Response: number analyzed (Participants) | 33
  First treatment - Complete Response + Partial Response | 69.7
  Second treatment - Complete Response + Partial Response | 0.0

11. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from start of treatment to death from any cause.
Time Frame: Duration of time from start of treatment to death from any cause. An average of 35.95 months.
Population: Analysis was performed for participants who underwent LAT in Cohorts 1 (n=13/24) and 2 (n=5/9) with initial Osimertinib start date as the start date of OS. Cohort 3 is not applicable for this outcome measure because these participants enrolled in the study after getting Osimertinib at an outside institution. One participant in Cohort 1 was not evaluable.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants in Cohort 1: Participants in Cohort 1 who underwent LAT.
- All Participants in Cohort 2: Participants in Cohort 2 who underwent LAT.
Arm/Group | All Participants in Cohort 1 | All Participants in Cohort 2
Number analyzed (Participants) | 13 | 5
Months | 38.2 [16.3 to 56.3] | 33.7 [18.5 to 40.3]

12. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as a Complete Response (CR) + Partial Response (PR) + Stable Disease (SD). Response was evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum diameters while on study. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progression.
Time Frame: end of treatment, up to 693 days
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 25 | 9 | 3
percentage of participants
  First Treatment - Complete Response + Partial Response + Stable Disease: number analyzed (Participants) | 25 | 9 | 0
  First Treatment - Complete Response + Partial Response + Stable Disease | 100 | 100 |
  Second Treatment - Complete Response + Partial Response + Stable Disease | 66.7 | 50.0 | 100

13. Secondary Outcome: Disease Control Rate (DCR) - All Participants
Description: as for outcome 12
Time Frame: end of treatment, up to 693 days
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | All Participants in Cohorts 1, 2, and 3
Number analyzed (Participants) | 36
percentage of participants
  First Treatment - Complete Response + Partial Response + Stable Disease: number analyzed (Participants) | 33
  First Treatment - Complete Response + Partial Response + Stable Disease | 100
  Second Treatment - Complete Response + Partial Response + Stable Disease | 66.7

14. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
Number analyzed (Participants) | 25 | 9 | 3
Participants | 25 | 9 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 74 months and 16 days, 65 months and 16 days, and 40 months and 4 days for the first, second and third group respectively.
Arm/Group | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib
All-Cause Mortality (participants affected / at risk) | 15/25 | 7/9 | 3/3
Serious Adverse Events (participants affected / at risk) | 14/25 | 5/9 | 2/3
Other Adverse Events (participants affected / at risk) | 24/25 | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer (N=25) | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation (N=9) | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, E. coli bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Inflenza A (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, Mental status change (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Myelitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysarthia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyrosine Kinase Inhibitor Naïve Epidermal Growth Factor Receptor *Mutated Non Small Cell Lung Cancer (N=25) | EGFR Mutated NSCLC Progressed on Prior 1st/2nd Generation EGFR TKI Therapy &Acquired T790M Mutation (N=9) | Epidermal Growth Factor Receptor Mutated Non Small Cell Lung Cancer Progressed on Osimertinib (N=3)
Abdominal pain (Gastrointestinal disorders) | 6 (10) | 3 (3) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (9) | 2 (2) | 1 (2)
Alkaline phosphatase increased (Investigations) | 3 (7) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (23) | 2 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (14) | 3 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 7 (7) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
CPK increased (Investigations) | 7 (23) | 2 (14) | 0 (0)
Cardiac disorders - Other, Atrial premature complex (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 3 (4) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (11) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (16) | 6 (10) | 1 (1)
Dizziness (Nervous system disorders) | 9 (11) | 4 (4) | 0 (0)
Dry eye (Eye disorders) | 5 (7) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (14) | 2 (4) | 2 (2)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 4 (5) | 0 (0)
Ear and labyrinth disorders - Other, Ear plugged (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, Muffled hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 2 (2) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (3) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 7 (13) | 7 (20) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Eye disorders - Other, CN 4 palsy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Diplopia (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (3)
Fatigue (General disorders) | 12 (18) | 4 (8) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 4 (9) | 2 (4) | 0 (0)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, Incision pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Loss of balance (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Sweating (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (11) | 4 (4) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8) | 2 (8) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (15) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (5) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Left thigh abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Viral pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, cold sore (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 9 (41) | 3 (6) | 2 (4)
Memory impairment (Nervous system disorders) | 3 (5) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, Muscle cramps (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (14) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Bilateral leg cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Bilateral calves cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (14) | 7 (10) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (33) | 1 (6) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (4) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 8 (16) | 5 (11) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (2) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 8 (9) | 3 (4) | 0 (0)
Paronychia (Infections and infestations) | 4 (5) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 7 (13) | 1 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 4 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Psychiatric disorders - Other, Erratic mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, Mental fog (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (26) | 2 (3) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hypoxemic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Shingles (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Serum amylase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (7) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Crack right and left thumb and left 3rd finger (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cracks around fingertips (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin lacerations (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, mild cracks at fingertips (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Incision site pain (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, abdominoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (3) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (7) | 2 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (5) | 2 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (15) | 2 (3) | 0 (0)
Watering eyes (Eye disorders) | 3 (4) | 1 (1) | 0 (0)
Weight loss (Investigations) | 10 (19) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
White blood cell decreased (Investigations) | 5 (32) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT02759835/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT02759835/ICF_001.pdf